CLINICAL TRIAL: NCT00687986
Title: A Randomized Clinical Trial of Surgery Versus Radiosurgery (Stereotactic Radiotherapy) in Patients With Stage IA NSCLC Who Are Fit to Undergo Primary Resection
Brief Title: Trial of Either Surgery or Stereotactic Radiotherapy for Early Stage (IA) Lung Cancer
Acronym: ROSEL
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, SSenan, Principal investigator, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ROSEL
Record Dates: First submitted 2008-05-28; First posted 2008-06-02 (Estimated); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Lung Cancer
Keywords: surgery; stereotactic radiotherapy; tumor control; quality of life
MeSH Terms: conditions — Lung Neoplasms | interventions — Radiosurgery; Radiotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- primary surgery (Active Comparator): primary surgical resection
  Interventions: Procedure: primary surgery
- stereotactic radiotherapy (Experimental): primary stereotactic radiotherapy
  Interventions: Radiation: stereotactic radiotherapy

INTERVENTIONS:
Radiation: stereotactic radiotherapy — Either 3 fractions of 20 Gray or 5 fractions of 12 Gy
  Other Names: radiotherapy
  Arms: stereotactic radiotherapy
Procedure: primary surgery — an anatomical surgical resection with lymph node dissection
  Other Names: operation
  Arms: primary surgery

SUMMARY:
The standard treatment for an early stage I lung cancer is surgery. However, surgery can be associated with complications and long-term impairment of the quality of life of patients. Stereotactic radiotherapy (SRT) is a outpatient technique which allows for local control rates that are comparable to those achieved using surgery. In this study, patients with stage IA non-small cell lung cancer will be randomized to either surgery or SRT in order to study the local and regional tumor control, quality of life and treatment costs at 2- and 5-years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a cytological or histological diagnosis of stage IA non-cell lung cancer diagnosed in accordance with Dutch CBO guidelines [2004]. When no pathological diagnosis is available, a patient with a new or growing pulmonary lesion with radiological features consistent with malignancy AND a lesion showing uptake on a FDG-PET scan will be eligible [Herder 2005].
* No evidence of regional or distant metastases on a standardized FDG-PET scan within 6 weeks of any protocol treatment .
* The medial extension of tumors should be least 2 cm away from main and lobar bronchi, and also minimum of 1.5 cm from large peripheral blood vessels such as the aorta and main pulmonary artery. Lesions of at least 2 cm from the mediastinal pleura will be eligible if the responsible radiation oncologist judges that the specified normal tissue tolerance doses specified in the protocol will not be exceeded.
* Patients who are judged by a multi-disciplinary team to have 2 primary lung tumors (on the basis of clinical, radiological, FDG-PET and/or cyto-pathology findings) are eligible for randomization provided that both surgery and SRT can be performed in accordance with protocol requirements.
* Patient should be fit to undergo a complete surgical resection of the lesion in accordance with Dutch CBO guidelines [2004]
* Performance score of ECOG ≤ 2 before any treatment.
* Able to comply with post-treatment follow-up
* Patients must sign and date a written Independent Ethics Committee approved informed consent form.

Exclusion Criteria:

* Prior chemotherapy or radiotherapy for the present diagnosis of NSCLC.
* History of any active malignancy (other than NSCLC) unless treated more than 3 years with curative intent and no recurrence, with the exception of non-melanoma skin cancers or in-situ cervical cancers.
* Any unstable systemic disease (including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, myocardial infarction within the previous year, severe cardiac arrhythmia requiring medication, hepatic, renal or metabolic disease).
* Concomitant treatment with any other experimental drug under investigation.
* Pregnancy
* Men and women of child-bearing potential not using effective means of contraception for 6 months after treatment has been completed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-10; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
local and regional control | 5 years

SECONDARY OUTCOMES:
Overall survival | 5 years
quality adjusted life years (QALYs) | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- VU University Medical Center, Amsterdam, Netherlands

REFERENCES:
- [Background] Haasbeek CJ, Senan S, Smit EF, Paul MA, Slotman BJ, Lagerwaard FJ. Critical review of nonsurgical treatment options for stage I non-small cell lung cancer. Oncologist. 2008 Mar;13(3):309-19. doi: 10.1634/theoncologist.2007-0195. PMID 18378542
- [Background] Hurkmans CW, Cuijpers JP, Lagerwaard FJ, Widder J, van der Heide UA, Schuring D, Senan S. Recommendations for implementing stereotactic radiotherapy in peripheral stage IA non-small cell lung cancer: report from the Quality Assurance Working Party of the randomised phase III ROSEL study. Radiat Oncol. 2009 Jan 12;4:1. doi: 10.1186/1748-717X-4-1. PMID 19138400
- [Background] Chang JY, Senan S, Paul MA, Mehran RJ, Louie AV, Balter P, Groen HJ, McRae SE, Widder J, Feng L, van den Borne BE, Munsell MF, Hurkmans C, Berry DA, van Werkhoven E, Kresl JJ, Dingemans AM, Dawood O, Haasbeek CJ, Carpenter LS, De Jaeger K, Komaki R, Slotman BJ, Smit EF, Roth JA. Stereotactic ablative radiotherapy versus lobectomy for operable stage I non-small-cell lung cancer: a pooled analysis of two randomised trials. Lancet Oncol. 2015 Jun;16(6):630-7. doi: 10.1016/S1470-2045(15)70168-3. Epub 2015 May 13. PMID 25981812
- [Background] Louie AV, van Werkhoven E, Chen H, Smit EF, Paul MA, Widder J, Groen HJ, van den Borne BE, De Jaeger K, Slotman BJ, Senan S. Patient reported outcomes following stereotactic ablative radiotherapy or surgery for stage IA non-small-cell lung cancer: Results from the ROSEL multicenter randomized trial. Radiother Oncol. 2015 Oct;117(1):44-8. doi: 10.1016/j.radonc.2015.08.011. PMID 26492839
- [Derived] Park S, Kim HJ, Park IK, Kim YT, Kang CH. Stereotactic ablative radiotherapy versus surgery in older patients with stage I lung cancer. Eur J Cardiothorac Surg. 2021 Jul 14;60(1):74-80. doi: 10.1093/ejcts/ezab045. PMID 33668061